CLINICAL TRIAL: NCT00694980
Title: A Phase I, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Intravenous and Subcutaneous rhuMAb Beta7 Administered in a Single-Dose, Dose-Escalation Stage Followed by a Multidose, Parallel-Treatment Stage in Patients With Ulcerative Colitis
Brief Title: A Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of rhuMAb Beta7 in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABS4262g; GA00930 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2008-06-07; First posted 2008-06-11 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Ulcerative Colitis
Keywords: UC; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: placebo; Drug: rhuMAb Beta7

INTERVENTIONS:
Drug: placebo — Intravenous and subcutaneous escalating doses
Drug: rhuMAb Beta7 — Intravenous and subcutaneous escalating doses

SUMMARY:
This is a randomized , double-blind, placebo-controlled study of approximately 70 patients with ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent
* 18-70 years of age
* Males and females with reproductive potential: Willing to use a reliable method of contraception
* Diagnosis of ulcerative colitis
* Eligible to receive biologic therapy
* Disease duration of >=12 weeks

Exclusion Criteria:

* Requirement for hospitalization due to severity of ulcerative colitis
* Moderate to severe anemia
* Any manifestation of ulcerative colitis or other conditions likely to require, in the investigator's judgment, treatment with >20 mg/day of prednisone, or prednisone equivalent, during the course of the study
* Pregnant or lactating
* Lack of peripheral venous access
* Inability to comply with study protocol
* History or presence of contraindicated diseases
* Congenital immune deficiency
* Active or prior infection with HIV or hepatitis B or C
* History of severe systemic bacterial, fungal, viral, or parasitic infections
* History of any other opportunistic infections within 12 weeks prior to initiation of study treatment
* Received a live attenuated vaccine within 4 weeks prior to screening
* Hospitalized within 4 weeks prior to screening
* Received any contraindicated therapy within 12 weeks prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of laboratory abnormalities | Through study completion or early study discontinuation
Incidence, nature, and severity of adverse events | Through study completion or early study discontinuation

SECONDARY OUTCOMES:
PK profile and parameters | Through study completion or early study discontinuation
Incidence of antibodies directed against rhuMAb Beta7 | Through study completion or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (28):
- United States (8):
  - Anniston, Alabama
  - San Francisco, California
  - Gainesville, Florida
  - Atlanta, Georgia
  - Lexington, Kentucky
  - Rochester, Minnesota
  - Great Neck, New York
  - Chapel Hill, North Carolina
- Leuven, Belgium
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - London, Ontario
  - Montreal, Quebec
- Germany (5):
  - Berlin
  - Frankfurt
  - Kiel
  - Regensburg
  - Ulm
- Netherlands (4):
  - Leiden
  - Maastricht
  - Nijmegen
  - Utrecht
- United Kingdom (4):
  - Bristol
  - London
  - Newcastle upon Tyne
  - Nottingham